CLINICAL TRIAL: NCT03133351
Title: Reference Range Analysis of the Entegrion Point of Care Coagulation Monitor (PCM™) in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Entegrion, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PCM-001
Record Dates: First submitted 2017-04-06; First posted 2017-04-28 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PCM: All enrolled subjects will have a blood sample tested using PCM.
  Interventions: Device: PCM

INTERVENTIONS:
Device: PCM — A fresh whole blood sample will be tested by PCM to determine the reference range.
  Other Names: Point of Care Coagulation Monitor

SUMMARY:
This study is intended to define the PCM normal laboratory range.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Body Mass Index (BMI) ≥ 19 and ≤ 30 kg/m2m with body weight ≥ 50 kg (106 lb)
3. Normal vital signs at screening

Exclusion Criteria:

1. Current daily tobacco use or previous recreational drug use
2. Pregnant or lactating at the time of the study
3. Currently taking any medications known to affect coagulation
4. History of excessive bleeding from minor trauma that required medical attention, spontaneous nose bleeds that required medical attention or multiple spontaneous abortions, liver disease, blood related diseases, congenital or acquired coagulopathies or thromboembolic diseases
5. Current diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 120 Males and 120 Females
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
PCM Clotting Time (CT) | Testing to be initiated within 4 minutes of sample collection
  To define the PCM normal laboratory reference range, PCM clotting time (CT) will be measured.
Clot Formation Time (CFT) | Testing to be initiated within 4 minutes of sample collection
  To define the PCM normal laboratory reference range, clot formation time (CFT) will be measured.
Alpha Angle (AA) | Testing to be initiated within 4 minutes of sample collection
  To define the PCM normal laboratory reference range, alpha angle (AA) will be measured.
  To define the PCM normal laboratory reference range, clot formation time (CFT) will be measured.
Maximum Clot Firmness (MCF) | Testing to be initiated within 4 minutes of sample collection
  To define the PCM normal laboratory reference range, maximum clot firmness (MCF) will be measured.
30-minutes Lysis after CT (LI30) | Testing to be initiated with 4 minutes of sample collection, with result available 30 minutes after CT
  To define the PCM normal laboratory reference range, 30-minutes lysis after CT (LI30) will be measured.
45-minutes Lysis after CT (LI45) | Testing to be initiated within 4 minutes of sample collection, with result available 45 minutes after CT
  To define the PCM normal laboratory reference range, 45-minutes lysis after CT (LI45) will be measured.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania